CLINICAL TRIAL: NCT00787943
Title: A Split-face, Paired-comparison, Pilot Study to Evaluate Safety and Efficacy of Two Topical Benzoyl Peroxide 10.0% Creams for Mild to Moderate Acne Vulgaris
Brief Title: Study of Two Different 10.0% Benzoyl Peroxide Creams for Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP-032408
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-03

CONDITIONS: Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left side of face (Experimental): Topical benzoyl peroxide 10.0% cream - Formulation 2 or Topical benzoyl peroxide 10.0% cream - Formulation 1 is to be applied to left side of the face.
  Interventions: Drug: Topical benzoyl peroxide 10.0% cream - Formulation 1; Drug: Topical benzoyl peroxide 10.0% cream - Formulation 2
- Right side of face (Experimental): Topical benzoyl peroxide 10.0% cream - Formulation 2 or Topical benzoyl peroxide 10.0% cream - Formulation 1 is to be applied to right side of the face.
  Interventions: Drug: Topical benzoyl peroxide 10.0% cream - Formulation 1; Drug: Topical benzoyl peroxide 10.0% cream - Formulation 2

INTERVENTIONS:
Drug: Topical benzoyl peroxide 10.0% cream - Formulation 1 — Formulation 1 will be applied to the randomly-assigned single (left or right) side of the face twice daily.
  Other Names: Benzoyl Peroxide 10% Cream
Drug: Topical benzoyl peroxide 10.0% cream - Formulation 2 — Formulation 1 will be applied to the randomly-assigned single (left or right) side of the face twice daily.
  Other Names: Benzoyl Peroxide 10% Cream

SUMMARY:
This study is a split face, paired-comparison, pilot study of 10 subjects. Participants in this study will be patients seen at Children's Memorial Hospital, who are clinically diagnosed with mild to moderate acne vulgaris. Participants will be recruited from the clinic, as well as advertising and from previous Institutional Review Board (IRB) approved acne studies housed in the Department of Dermatology. All subjects accrued from previous studies have agreed to be contacted for further investigations. Subjects 13 to 35 years of age with mild to moderate acne vulgaris symmetrical in appearance on both sides of the face, and meeting inclusion criteria will be eligible to participate.

DETAILED DESCRIPTION:
Acne vulgaris is a follicular disorder occurring in pilosebaceous units in the skin of the face, neck, and upper trunk. These sebaceous follicles have follicular channels and adjacent multiacinar sebaceous glands. In the lubrication process of normal skin, sebum travels through the follicular canal to the skin surface, carrying along with it desquamated cells from follicular epithelium. Acne develops when these specialized follicles undergo pathologic alterations that result in the formation of non-inflammatory lesions (comedones) and inflammatory lesions (papules, pustules, and nodules).

The basic cause of acne remains unknown, but its manifestations are thought to be the product of four pathogenic events: 1) increased sebum production fueled by androgenic stimulation in the pubertal period; 2) obstruction of the pilosebaceous unit due to an abnormal keratinization process; 3) proliferation of Propionibacterium acnes, an anaerobic diptheroid normally residing in pilosebaceous follicles; and 4) inflammation that is mediated both by the action of chemotactic factors and various enzymes, and initiated in part by the interaction of P. acnes with toll-like receptors. Impaction of the pilosebaceous follicle gives rise to the microcomedo that is thought to be the precursor lesion of acne.

Topical benzoyl peroxide is a common and well-established agent with known antibacterial and antimicrobial properties used in the treatment of acne vulgaris. The safety profile for topical benzoyl peroxide has been well delineated. The most common side effects attributed to benzoyl peroxide products include irritation, dryness, scaling, burning and stinging.

Benzoyl peroxide 10.0% creams (Formulation #1 and Formulation #2) will be evaluated to detect any differences in their response for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects who are 13 to 35 years of age.
2. Subjects are in good health and are free of any other facial skin disorders that may interfere with acne study assessments.
3. Subjects have the willingness and ability to understand and provide informed assent/consent to participate in the study and are able to communicate with the investigator. Subjects are willing and able to follow all study directions and to commit to all follow-up visits for the duration of the study. In addition, subjects must be willing to accept the restrictions of the study.
4. A minimum of 5 inflammatory lesions (papules and pustules) on each side of the face, and a minimum of 5 non-inflammatory lesions (open comedones and closed comedones) on each side of the face. Lesions should be relatively symmetrical in appearance on both sides of the face. At least one inflammatory lesion should be measured no smaller than 2 mm in diameter and should be visible on each side of the face in images taken with digital imaging station.
5. Ongoing oral medications (other than those specifically for acne) are acceptable provided subjects are on a stable regimen throughout the study and provided the medications are determined likely to not interfere with study assessments.
6. Subjects will not use medicated cosmetics and/or soaps (including soaps containing antibacterial agents such as benzoyl peroxide, keratolytic agents such as salicylic acid, skin fresheners/astringents or aftershave lotions) for the duration of the study.
7. Subjects who agree not to use any other acne treatment (including prescription and non-prescription medications) on the test site for the duration of the study.
8. Subjects who agree not to change facial cosmetic products during the study.
9. Subjects who agree to only use sunscreen/sunblock agents that are labeled as non-comedogenic.

Exclusion Criteria:

1. Subjects or parents of subjects who are unable to understand the protocol or to give informed consent/assent.
2. Subjects with mental illness.
3. Subjects with no inflammatory acne.
4. Subjects with any acne cysts or nodules.
5. Subjects with acne conglobata, acne fulminans, secondary acne (e.g. Chloracne, drug-induced acne), or any acne requiring systemic treatment.
6. Subjects with excessive facial hair that may interfere with study assessments.
7. Subjects with other facial skin disorders that may interfere with study assessments.
8. Subjects with a history of skin cancer or actinic keratosis.
9. Subjects who have used tanning devices within one week prior to baseline study visit.
10. Subjects who have applied any topical products (e.g. emollients, sunscreens) or any cosmetics to the face at least one hour prior to study assessments.
11. Use of hormonal oral contraceptives for acne control or for less than 6 months prior to study baseline.
12. Subjects with known allergies, a history of allergy or sensitivity to benzoyl peroxide, or any of the test article components.
13. Subjects using topical or systemic medication within 14 days before the study entry, which could interfere with study assessments. This includes but is not limited to the following: anti-inflammatory drugs (e.g. topical and systemic corticosteroids and systemic antihistamines), anti-acne drugs, topical and oral retinoids, topical antibacterial agents to the face, and any immunosuppressive drugs. Ongoing oral medications not expected to interfere with study assessments are allowed if the subject is on a stable regimen.
14. Subjects who are currently enrolled in another clinical investigation or have been enrolled in an acne trial within a period of 30 days prior to enrollment in this study.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the clinic, as well as advertising in the Department of Dermatology.
Groups:
- All Study Participants: Apply Formula #1 to assigned side of face twice daily. Apply Formula #2 to assigned side of face twice daily.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Inflammatory Lesions (Papules and Pustules)
Description: Assessment will be done based on lesion counting. We will compare the lesions treated twice daily with the benzoyl peroxide 10.0% cream Formulation #1 vs. the benzoyl peroxide 10.0% cream Formulation #2.
Time Frame: 4 Weeks
Population: Papules and pustules were analyzed on the left and right side of the face for each of the 10 subjects. Analysis was per protocol with intention to treat.
Measure: Number; unit: Lesions
Groups:
- Papules: Benzoyl Peroxide 10.0% Cream Formulation #1; Pustules: Benzoyl Peroxide 10.0% Cream Formulation #1; Papules: Benzoyl Peroxide 10.0% Cream Formulation #2; Pustules: Benzoyl Peroxide 10.0% Cream Formulation #2: Apply a pea size amount two times a day, in the morning and evening. Smooth evenly into skin until it becomes invisible.
Arm/Group | Papules: Benzoyl Peroxide 10.0% Cream Formulation #1 | Pustules: Benzoyl Peroxide 10.0% Cream Formulation #1 | Papules: Benzoyl Peroxide 10.0% Cream Formulation #2 | Pustules: Benzoyl Peroxide 10.0% Cream Formulation #2
Number analyzed (Participants) | 10 | 10 | 10 | 10
Lesions
  Subject 1 Day 0 | 6 | 3 | 10 | 0
  Subject 1 Day 2 | 1 | 0 | 5 | 1
  Subject 1 Day 7 | 1 | 0 | 1 | 0
  Subject 1 Day 28 | 6 | 1 | 4 | 2
  Subject 2 Day 0 | 14 | 2 | 7 | 0
  Subject 2 Day 2 | 15 | 1 | 12 | 2
  Subject 2 Day 7 | 7 | 0 | 4 | 0
  Subject 2 Day 28 | 7 | 0 | 8 | 9
  Subject 3 Day 0 | 7 | 0 | 9 | 6
  Subject 3 Day 2 | 8 | 0 | 7 | 0
  Subject 3 Day 7 | 5 | 3 | 11 | 1
  Subject 3 Day 28 | 8 | 0 | 0 | 1
  Subject 4 Day 0 | 14 | 4 | 6 | 1
  Subject 4 Day 2 | 20 | 1 | 4 | 1
  Subject 4 Day 7 | 21 | 0 | 7 | 1
  Subject 4 Day 28 | 10 | 1 | 9 | 1
  Subject 5 Day 0 | 23 | 1 | 23 | 2
  Subject 5 Day 2 | 26 | 18 | 28 | 21
  Subject 5 Day 7 | 31 | 0 | 31 | 4
  Subject 5 Day 28 | 26 | 1 | 29 | 2
  Subject 6 Day 0 | 22 | 2 | 6 | 3
  Subject 6 Day 2 | 14 | 0 | 6 | 2
  Subject 6 Day 7 | 10 | 1 | 10 | 1
  Subject 6 Day 28 | 12 | 1 | 11 | 0
  Subject 7 Day 0 | 34 | 6 | 30 | 5
  Subject 7 Day 2 | 47 | 3 | 34 | 7
  Subject 7 Day 7 | 46 | 3 | 53 | 1
  Subject 7 Day 28 | 35 | 6 | 33 | 4
  Subject 8 Day 0 | 9 | 1 | 7 | 1
  Subject 8 Day 2 | 11 | 0 | 5 | 0
  Subject 8 Day 7 | 10 | 0 | 3 | 0
  Subject 8 Day 28 | 6 | 0 | 7 | 0
  Subject 9 Day 0 | 17 | 1 | 19 | 1
  Subject 9 Day 2 | 21 | 0 | 19 | 0
  Subject 9 Day 7 | 22 | 0 | 14 | 0
  Subject 9 Day 28 | 13 | 0 | 11 | 0
  Subject 10 Day 0 | 13 | 2 | 13 | 4
  Subject 10 Day 2 | 15 | 0 | 18 | 1
  Subject 10 Day 7 | 13 | 1 | 7 | 2
  Subject 10 Day 28 | 6 | 1 | 9 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Benzoyl Peroxide 10.0% Cream Formulation #1: Formulation #1 applied to one side of the face by all 10 subjects.
- Benzoyl Peroxide 10.0% Cream: Formulation #2: Formulation #2 applied to one side of the face by all 10 subjects.
Arm/Group | Benzoyl Peroxide 10.0% Cream Formulation #1 | Benzoyl Peroxide 10.0% Cream: Formulation #2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benzoyl Peroxide 10.0% Cream Formulation #1 (N=10) | Benzoyl Peroxide 10.0% Cream: Formulation #2 (N=10)
Burning/Stinging (Skin and subcutaneous tissue disorders) | 8 (40) | 8 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No